CLINICAL TRIAL: NCT01055249
Title: Single Centre, Subject and Observer Blinded, Placebo Controlled, Cross-over Study of the Effect of Oral Ibuprofen and Topical Hydrocortisone-21-acetate on Ultraviolet Radiation (UVR) Induced Pain and Inflammation in Healthy Volunteers
Brief Title: UVB Model Validation Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X-pert Med GmbH (Industry)
Responsible Party: Ilka Rother, MD, X-pert Med GmbH
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: XPM-024
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Pain; Inflammation; Healthy Volunteers
Keywords: UVB; pain; inflammation; model; healthy volunteers; Ultraviolet radiation (UVR) induced pain and inflammation in healthy volunteers
MeSH Terms: conditions — Pain; Inflammation | interventions — Ibuprofen; Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Ibuprofen 600 mg (active comparator); Hydrocortisone 15 microl/cm2 (active comparator); Placebo Gel (placebo comparator)
  Interventions: Drug: Ibuprofen, Hydrocortisone
- Group B (Other): Oral Placebo (placebo comparator), Hydrocortisone 15 microl/cm2 (active comparator); Placebo Gel (placebo comparator)
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Ibuprofen, Hydrocortisone — Ibuprofen 600 mg film coated tablets, b.i.d., Hydrocortisone-21-acetate creme (25%) 15 microl/cm2 b.i.d.
  Arms: Group A
Drug: Hydrocortisone — Hydrocortisone-21-acetate creme (25%) 15 microl/cm2 b.i.d.
  Arms: Group B

SUMMARY:
Single centre, subject and observer blinded, placebo controlled, cross-over study of the effect of oral ibuprofen and topical hydrocortisone-21-acetate on ultraviolet radiation (UVR) induced pain and inflammation in healthy volunteers conducted in two segments and using an intra-individual comparison of application areas.

DETAILED DESCRIPTION:
Single centre, subject and observer blinded, placebo controlled, cross-over study of the effect of oral ibuprofen and topical hydrocortisone-21-acetate on ultraviolet radiation (UVR) induced pain and inflammation in healthy volunteers conducted in two segments and using an intra-individual comparison of application areas.

Subjects that signed the informed consent and are eligible to the study will be irradiated on the back to evaluate their individual minimal erythema doses (MEDs). Read out to determine MED will be done within 24 h after UVR.

A training session (without study medication) using the MED definition areas will be performed in order to introduce subjects to the testing and rating procedures.

Subjects will come in within 14 days of screening to start the first Segment of the study. Eligible subjects will be randomised to receive either:

1. IB 600 mg, applied orally b.i.d., or
2. OP, applied orally b.i.d.

Allocation of topical treatment to these areas will be randomly assigned to:

1. PG, 15 μl/cm2 applied topically b.i.d., or
2. HC, 15 μl/cm2 applied topically b.i.d.

Defined areas will be irradiated with defined dosages of UVR. Assessment of hyperalgesia to heat and signs of inflammation (erythema, skin temperature) for all areas will be performed.

Subjects return within 4 to 11 days to the study site for the second segment of the study. Treatment allocation will be crossed-over and new treatment areas will be selected on the back.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

-

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Hyperalgesia to heat | 72 h

SECONDARY OUTCOMES:
Erythema, Skin temperature | 72 h

CONTACTS AND LOCATIONS:
Locations (1):
- X-pert Med GmbH, Gräfelfing, Bavaria, Germany